CLINICAL TRIAL: NCT06664021
Title: Exploring the Efficacy and Safety of Tislelizumab in Combination With S-1 in the Treatment of Patients With Postoperative Recurrent High-risk Intrahepatic Cholangiocarcinoma：A Prospective, Multicenter, Phase II Clinical Study
Brief Title: Exploring the Efficacy and Safety of Tislelizumab in Combination With S-1 in the Treatment of Patients With Postoperative Recurrent High-risk Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024KY467
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Tislelizumab + S-1
  Interventions: Drug: Tislelizumab combined with S-1
- No treatment group (No Intervention): No postoperative adjuvant therapy is performed

INTERVENTIONS:
Drug: Tislelizumab combined with S-1 — Tislelizumab：200mg q3w iv , lasts for one year. S-1：40mg, 50mg, or 60mg orally twice daily for 4 weeks, depending on body surface area, followed by 2 weeks of rest，lasts four cycles.
  Arms: Treatment group

SUMMARY:
Evaluating the efficacy and safety of treatment with Tislelizumab in combination with S-1 in patients with high-risk recurrent intrahepatic cholangiocarcinoma after radical surgery

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old, male and female;
* Intrahepatic cholangiocarcinoma was pathologically confirmed after R0 or R1 resection. Patients were also pathologically confirmed to have one of the following high-risk factors (i.e., positive margins, multiple tumor nodes, positive lymph nodes, positive perineural infiltration, intrahepatic cholangiocarcinoma >5 cm in diameter, and combined vascular invasion);
* Enhanced computed tomography (CT) scans of the chest, abdomen, and pelvis were required within 30 days prior to surgery to demonstrate the absence of distant tumor metastases;
* No history of any chemotherapy, radiotherapy, immunotherapy or interventional therapy within 3 months prior to surgical resection;
* Child-Pugh grade A or B, ECOG score 0-1;
* Normal organ function prior to drug administration: ANC ≥1.5×10^9/L, Hemoglobin ≥90g/L, PLT >50*10^9/L, serum creatinine (SCr) ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥50 ml/min (Cockcroft-Gault formula); total bilirubin (TBIL) ≤2 times the upper limit of normal (ULN); glutamine transaminase (AST) or glutamine transaminase (ALT) levels ≤3 times the ULN; urinary protein <2+ (if urinary protein) upper limit of normal (ULN); albumin transaminase (AST) or alanine transaminase (ALT) levels ≤3 times upper limit of normal (ULN); urine protein <2+ (if urine protein ≥2+, 24-hour urine protein quantification must show ≤1g of protein); and adequate surgical biliary drainage with no signs of infection.
* Normal coagulation function: a. International normalized ratio INR ≤ 1.5 x ULN; b. Partial thromboplastin time APTT ≤ 1.5 x ULN; c. Prothrombin time PT ≤ 1.5 ULN;
* In case of hepatitis B virus (HBV) infection: if HBsAg-positive, HBV-DNA testing is required and HBV-DNA must be <2000 IU/mL and willing to receive antiviral therapy throughout the study period; hepatitis C virus (HCV)-RNA-positive patients must have HCV-RNA <1×10^3copy/mL and must receive antiviral therapy according to treatment guidelines.
* No major abnormalities in heart, lung or kidney function;
* No history of gastrointestinal hemorrhage;
* Sign the informed consent form.

Exclusion Criteria:

* The tumor is not completely resected, or the pathological diagnosis suggests non-intrahepatic cholangiocarcinoma such as hepatocellular carcinoma, mixed hepatocellular carcinoma, and hepatoportal cholangiocarcinoma;
* Pregnant or breastfeeding women;
* Combined with other malignant tumors;
* Have any active autoimmune disease or a history of autoimmune disease;
* Uncontrolled clinically significant cardiac disease, including but not limited to the following: (1) > NYHA II congestive heart failure; (2) unstable angina pectoris; (3) myocardial infarction within the last 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention;
* The patient has a congenital or acquired immunodeficiency;
* Uncontrollable infection > grade 2 (NCI-CTC version 5.0);
* Psychopaths;
* Patients have participated in other clinical trials within the past three months;
* Postoperative patients receiving other targeted agents, immunotherapy such as PD-1 antibodies, and FOLFOX systemic chemotherapy;
* Patients who are not suitable to participate in the study as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-16 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
1-year RFS rate | 12 months
  Proportion of patients with no local, regional, or metastatic ICC or death from any cause (whichever occurs first) 12 months after hepatectomy.

SECONDARY OUTCOMES:
RFS | 24 months
  Time from hepatectomy to the first documented occurrence of local, regional, or metastatic ICC or death from any cause, whichever occurs first.
OS | 24 months
  Time from hepatectomy to first recorded occurrence of death from any cause
Survival time after recurrence | 24 months
  The time from the first documented occurrence of localized, regional, or metastatic ICC, whichever occurs first, to death from any cause.
AEs AEs AEs AEs AE | 24 months
  Adverse Events (AEs)The grade of AEs and the number of patients with AEs are assessed based on CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Lian-xin Liu, Principal Investigator — Anhui Provincial Hospital
Locations (2):
- China (2):
  - No.2 People's Hospital of Fuyang city, Fuyang, Anhui
  - Anhui province hospital, Hefei, Anhui

IPD SHARING:
Plan to Share IPD: No